CLINICAL TRIAL: NCT05980000
Title: Open-Label, Randomized Phase 2 Trial of Ramucirumab in Combination With Pembrolizumab Versus Pembrolizumab Alone as First-Line Treatment of PD-L1 Positive, Recurrent or Metastatic Head and Neck Squamous-Cell Carcinoma (RM-HNSCC)
Brief Title: Ramucirumab and Pembrolizumab vs Pembrolizumab Monotherapy in PD-L1 Positive Head and Neck Squamous-Cell Carcinoma
Acronym: Rambro2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202308161
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Head and Neck Cancer; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Carcinoma; Metastatic Head-and-neck Squamous-cell Carcinoma; Metastatic Head and Neck Cancer; HNSCC
Keywords: PD-L1 positive RM-HNSCC; RM-HNSCC; oral cavity HNSCC; oropharynx HNSCC; larynx HNSCC; hypopharynx HNSCC
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Ramucirumab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomized on a 2:1 basis to Arm 1 or Arm 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: Ramucirumab and Pembrolizumab (Experimental): Patients receive ramucirumab IV and pembrolizumab IV every 3 weeks. Cycles are 21 days in length. Treatment will continue until progression or unacceptable toxicity for up to 35 cycles of treatment.
  Interventions: Drug: Ramucirumab; Drug: Pembrolizumab
- Arm 2: Pembrolizumab monotherapy (Active Comparator): Patients receive pembrolizumab IV every 3 weeks. Cycles are 21 days in length. Treatment will continue until progression or unacceptable toxicity for up to 35 cycles of treatment.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Ramucirumab — Ramucirumab is administered at a dose of 10 mg/kg over 60 minutes.
  Other Names: Cyramza
  Arms: Arm 1: Ramucirumab and Pembrolizumab
Drug: Pembrolizumab — Pembrolizumab is administered at a flat dose of 200 mg over 30 minutes.
  Other Names: MK-3475; Keytruda

SUMMARY:
This is a phase 2 study investigating the efficacy of ramucirumab in combination with pembrolizumab compared to pembrolizumab monotherapy. Ramucirumab is a VEGFR-2 inhibitor believed to potentially enhance the efficacy of PD-1 inhibitors such as pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Incurable RM-HNSCC, defined as RM disease or second or subsequent primary HNSCC not amenable to cure by surgery and/or radiation therapy or patient declines or is ineligible for curative therapy. Eligible primary tumor sub-sites include oral cavity, oropharynx, larynx and hypopharynx only.
* PD-L1 positive (CPS ≥1) disease, based on local IHC assay using 22C3 antibody.
* Measurable disease per RECIST 1.1.
* No prior systemic therapy for RM-HNSCC. RM disease developing within 6 months of completion of either a) systemic platinum or cetuximab therapy given as a component of a curative-intent multi-modality regimen or b) radiation therapy and/or surgery is eligible.
* At least 18 years of age.
* ECOG performance status 0-1.
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN. In the setting of liver metastases, AST(SGOT)/ALT(SGPT) ≤ 5.0 x IULN
  * Creatinine ≤ 1.5 x ULN. If patient has creatinine > 1.5 x ULN, then 24 hour urine collection must be performed and creatinine clearance must be ≥ 40 mL/min by Cockcroft-Gault
  * Urine protein to creatinine ratio (UPC) ≤ 1; if UPC > 1, then a 24-hour urine protein must be assessed and patient must have a 24-hour urine protein value < 1 g to be eligible
  * INR ≤ 1.5 (≤ 3.0 if on warfarin) and PTT ≤ 1.5 x ULN (Patients are allowed to be on anticoagulation)
* The effects of Ramucirumab on the developing human fetus are unknown. For this reason and because VEGFR2 inhibiting agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 28 days after completion of the study.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* PD-L1 negative (CPS 0) disease, based on local IHC assay using 22C3 antibody.
* Cutaneous or nasopharynx SCC.
* Major surgery within 28 days prior to C1D1, minor surgery or subcutaneous venous access device placement within 7 days prior to C1D1, history of significant tumor site bleeding within 14 days prior to C1D1, or elective or planned major surgery to be performed during the course of the clinical trial.
* Palliative radiation therapy within 2 weeks of C1D1.
* Serious or non-healing, non-malignant wound, ulcer, or bone fracture within 28 days prior to C1D1.
* A history of other malignancy ≤ 1 year previous with the exception of completely resected skin carcinoma or other cancers with a low risk (<10%) of recurrence over the next 2 years.
* Cirrhosis at a level of Child-Pugh B (or worse). Cirrhosis of any degree with a history of hepatic encephalopathy or clinically meaningful ascites (from cirrhosis requiring diuretics or paracentesis).
* Currently receiving any other investigational agents.
* Ongoing toxicity attributed to prior anti-cancer therapy that is > grade 1, except alopecia, anemia, lymphopenia, xerostomia, fatigue or rash.
* Active central nervous system metastases: defined as currently receiving radiation therapy to metastatic CNS disease. Once radiation therapy is completed and patient has completed a 2 week washout, patients with CNS disease are eligible if they meet all other criteria for enrollment.
* A history of severe allergic reactions attributed to compounds of similar chemical or biologic composition to Ramucirumab or other agents used in the study.
* Serious uncontrolled intercurrent illness within the 3 months prior to study entry including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, or cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving systemic corticosteroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of intense immunosuppressive therapy within 7 days prior to C1D1.
* Active autoimmune disease (i.e. rheumatoid arthritis, lupus) that has required IV or subcutaneous systemic treatment in the past 6 months prior to C1D1 (excluding Rituxan). Replacement therapy (i.e. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* GI perforation or fistula within 6 months of C1D1. Malignant oral fistulas are not excluded.
* History of inflammatory bowel disease, ulcerative colitis, or Crohn's disease.
* Poorly controlled hypertension (defined as serial high blood pressure measurements [systolic blood pressures of > 160 mmHg or diastolic blood pressures of > 100 mmHg] documented during the four-week interval prior to C1D1) despite standard medical management. Initiation or adjustment of antihypertensive medications to control blood pressure is permitted prior to study entry.
* Arterial thromboembolic events (including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina) within 6 months, prior to C1D1.
* Deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") within 3 months prior to C1D1.
* Any bleeding (grade 3 or 4) within 3 months prior to C1D1.
* Receiving chronic antiplatelet therapy, including nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
* Current, active bleeding (within 14 days prior to C1D1) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices), if patients are taking an oral anticoagulant or low molecular weight heparin. Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or LMWH prior to C1D1.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From start of study treatment through completion of treatment (estimated to be 24 months)
  ORR is defined as the number of patients with a complete response (CR) and a partial response (PR) by RECIST 1.1 criteria. A CR is defined as the disappearance of all target lesions, reduction in pathological lymph nodes to <10 mm in short axis, and disappearance of all non-target lesions with normalization of tumor marker level. A PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Duration of Response (DoR) | From time criteria is met for CR or PR through completion of treatment (estimated to be 1 year and 40 weeks)
  Duration of overall response is measured from the time criteria are met for a CR or PR per RECIST 1.1 (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Duration of overall CR is measured from the time criteria are met for a CR per RECIST 1.1 until the first date that progressive disease is objectively documented.
Progression-Free Survival (PFS) | From start of study treatment through 5 years
  PFS is defined as the duration of time from the start of treatment to time of progression or death, whichever occurs first.
Overall Survival (OS) | From start of study treatment through 5 years
  OS is defined as the time from start of treatment to the date of death, censored at the last follow-up otherwise.
Incidence rate, frequency, and severity of adverse events (AEs) | From start of study treatment through 30 days after last dose (expected to be 2 years and 1 month)
  AEs will be assessed using CTCAE v4.0 and summarized by arm.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu